CLINICAL TRIAL: NCT06470386
Title: The Efficacy and Safety of Compound Alverine Citrate Soft Capsules in the Treatment of Portal Hypertension in Patients With Liver Cirrhosis: a Prospective, Open-label, Multicentre, Randomised Controlled Trial
Brief Title: The Efficacy and Safety of Alverine in the Treatment of Portal Hypertension in Patients With Liver Cirrhosis
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Shandong Provincial Hospital (Other Government); Shanghai East Hospital (Other); Shanghai Zhongshan Hospital (Other); Affiliated Drum Tower Hospital of Nanjing University Medical School (Unknown); The First Affiliated Hospital of Nanchang University (Other); Shanghai Public Health Clinical Center (Other Government); Daping Hospital, Army Medical Center of PLA (Other)
Responsible Party: Principal Investigator, Wei-Fen Xie, Director, Department of Gastroenterology, Changzheng Hospital, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZXH-PH-ALV-2401
Record Dates: First submitted 2024-06-11; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Hypertension, Portal
Keywords: Cirrhotic portal hypertension; Alverine; Pharmacological therapy
MeSH Terms: conditions — Hypertension, Portal | interventions — alverine; Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alverine Group (Experimental): Compound Alverine Citrate Capsules (Lejiansu; specification: each capsule contains 60 mg of Alverine Citrate and 300 mg of Simethicone; manufactured by the French company UCB Pharma), 180 mg/day (1 capsule orally, 3 times a day), taken continuously for 24 weeks.
  Interventions: Drug: Alverine
- Carvedilol Group (Active Comparator): Jinluo (Carvedilol Tablets; specification: 6.25 mg; manufactured by Qilu Pharmaceutical Co., Ltd.), taken orally, starting dose of 6.25 mg once a day, gradually adjusted according to heart rate to 6.25 mg twice a day, 12.5 mg in the morning and 6.25 mg in the evening, 12.5 mg twice a day, or adjusted to the maximum tolerated dose (heart rate greater than 55 beats/min and systolic blood pressure greater than 90 mmHg), taken continuously for 24 weeks.
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Alverine — 180 mg/day (1 capsule orally, 3 times a day), taken continuously for 24 weeks
  Other Names: Compound Alverine Citrate Capsules
  Arms: Alverine Group
Drug: Carvedilol — taken orally, starting dose of 6.25 mg once a day, gradually adjusted according to heart rate to 6.25 mg twice a day, 12.5 mg in the morning and 6.25 mg in the evening, 12.5 mg twice a day, or adjusted to the maximum tolerated dose (heart rate greater than 55 beats/min and systolic blood pressure greater than 90 mmHg), taken continuously for 24 weeks.
  Other Names: Jinluo
  Arms: Carvedilol Group

SUMMARY:
Study Overall Design:

This trial is a prospective, open-label, multicenter, randomized controlled clinical trial. Subjects who meet the inclusion criteria and do not meet the exclusion criteria will be randomly assigned to either the Alverine treatment group or the Carvedilol treatment group in a 1:1 ratio after signing the informed consent form. After randomization, participants will enter a 24-week medication period. Apart from the baseline period, the efficacy of the treatment will be evaluated 24 weeks post-treatment. The safety evaluation will be conducted according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 by the National Cancer Institute.

Study Population:

Patients with cirrhotic portal hypertension.

Interventions:

Alverine Group: Compound Alverine Citrate Capsules (Lejiansu; each capsule contains 60 mg of Alverine Citrate and 300 mg of Simethicone; manufactured by the French company UCB Pharma), 180 mg/day (1 capsule orally, 3 times a day), taken continuously for 24 weeks.

Carvedilol Group: Jinluo (Carvedilol Tablets; 6.25 mg; manufactured by Qilu Pharmaceutical Co., Ltd.), taken orally, starting dose of 6.25 mg once a day, gradually adjusted according to heart rate to 6.25 mg twice a day, 12.5 mg in the morning and 6.25 mg in the evening, 12.5 mg twice a day, or adjusted to the maximum tolerated dose (heart rate greater than 55 beats/min and systolic blood pressure greater than 90 mmHg), taken continuously for 24 weeks.

Study Objectives:

1. Primary Study Objective Evaluate the efficacy and safety of Compound Alverine Citrate Capsules in the treatment of cirrhotic portal hypertension.
2. Secondary Study Objectives Evaluate the effect of Compound Alverine Citrate Capsules on the incidence of esophagogastric variceal bleeding and other cirrhotic decompensation events.
3. Exploratory Study Objectives Evaluate the efficacy of Compound Alverine Citrate Capsules in the treatment of cirrhotic portal hypertension using other non-invasive detection methods. Observe the effects of Compound Alverine Citrate Capsules on the multi-omics characteristics of cirrhosis, reversal of portal hypertension, recompensation of decompensated cirrhosis, and prevention of the progression of cirrhosis to liver cancer.

Study Endpoints:

(1) Primary Study Endpoints

1. The treatment response rate, defined as a reduction in HVPG of ≥10% from baseline or a reduction to below 12 mmHg after 24 weeks of treatment.
2. The incidence, events, and severity of adverse events, serious adverse events, and adverse events leading to treatment discontinuation after treatment (evaluated according to CTCAE version 5.0).

(2) Secondary Study Endpoints

1. Incidence of esophagogastric variceal bleeding during treatment.
2. Incidence of other cirrhotic decompensation events (new onset or progression of ascites, spontaneous bacterial peritonitis, overt hepatic encephalopathy, acute kidney injury/hepatorenal syndrome, primary liver cancer, etc.) during treatment.
3. Reduction in HVPG from baseline after 24 weeks of treatment.
4. Mortality/liver transplantation rate during treatment.
5. Overall survival time of subjects.
6. Reduction in mean arterial pressure (MAP) and heart rate from baseline after 24 weeks of treatment.

(3) Exploratory Study Endpoints

1. Changes in liver stiffness and spleen stiffness from baseline after 24 weeks of treatment.
2. Improvement in liver function (Child-Pugh score, MELD score) after 24 weeks of treatment.
3. Changes in cardiac function (left ventricular ejection fraction) from baseline after 24 weeks of treatment.
4. Changes in imaging characteristics, blood/stool metabolomics characteristics, portal hypertension reversal biomarkers, cirrhosis recompensation biomarkers, and cirrhosis progression to liver cancer biomarkers after 24 weeks of treatment.

Sample Size Calculation:

In animal experiments, it was confirmed that there was no statistically significant difference in the effect of Alverine and Carvedilol in treating portal hypertension. Literature reports indicate that the treatment response rate of Carvedilol for cirrhotic portal hypertension is approximately 60%. Based on the sample size calculation method for non-inferiority trials with two samples, with a non-inferiority margin δ=0.20, a one-sided α=0.025, and β=0.2, the calculated sample size for each group is 74 cases, totaling 148 cases. Considering a 20% dropout rate, a total of 178 cases are needed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80 years (inclusive), regardless of gender.
2. Patients with cirrhosis confirmed by clinical, laboratory, imaging examinations, and/or liver biopsy.
3. Hepatic venous pressure gradient (HVPG) ≥ 10 mmHg.
4. Agree to participate and sign the informed consent form.

Exclusion Criteria:

1. Use of non-selective beta-blockers such as Carvedilol, Propranolol, or Alverine, Papaverine, and their derivatives (e.g., Papaverine Hydrochloride, Drotaverine Hydrochloride) within 4 weeks prior to enrollment.
2. Previous surgeries including transjugular intrahepatic portosystemic shunt (TIPS) or liver transplantation.
3. History or current occurrence of overt hepatic encephalopathy, esophagogastric variceal bleeding, or grade 3 ascites.
4. Use of vasoactive drugs such as somatostatin and its analogs, vasopressin, terlipressin, dopamine, norepinephrine within 1 week prior to enrollment.
5. History of heavy alcohol consumption within 12 weeks prior to enrollment and inability to abstain from heavy drinking during the study (equivalent to ethanol intake ≥30 g/day for males, ≥20 g/day for females).
6. Serum total bilirubin level ≥3×ULN (≥5×ULN for autoimmune liver disease patients), or serum sodium level <125 mmol/L, or white blood cell count <1×10^9/L, or platelet count <30×10^9/L, or International Normalized Ratio (INR) >2.3.
7. Significant renal insufficiency (eGFR (CKD-EPI formula) <20 mL/min/1.73 m²).
8. Presence of thrombosis or cavernous transformation in the portal venous system (including portal vein, splenic vein, superior mesenteric vein); patients with a history of portal vein thrombosis can be enrolled if no definite thrombosis is detected in the portal venous system within 2 weeks.
9. HBV DNA or HCV RNA > the lower limit of detection; patients with active HCV antiviral treatment; patients on anti-HBV treatment for less than 24 weeks.
10. Uncontrollable active infections (such as lung infection, abdominal infection, HIV, etc.) within 4 weeks prior to enrollment.
11. Poorly controlled hypertension, diabetes, or other severe heart or lung diseases.
12. Diagnosed or suspected malignancies, including liver cancer.
13. Known allergy to Alverine, Papaverine and their derivatives (e.g., Papaverine Hydrochloride, Drotaverine Hydrochloride) or Carvedilol; contraindications for Carvedilol: NYHA class IV decompensated heart failure requiring intravenous inotropic drugs; asthma, chronic obstructive pulmonary disease (COPD) with bronchospasm; second or third degree atrioventricular block, severe bradycardia (heart rate less than 50 bpm), sick sinus syndrome (including sinoatrial block); cardiogenic shock; severe hypotension (systolic blood pressure less than 85 mmHg).
14. Patients with glaucoma.
15. Patients with psychiatric disorders.
16. Pregnant or lactating women, or women with potential for pregnancy.
17. Participation in other drug trials within 4 weeks prior to enrollment.
18. Other reasons deemed unsuitable by the researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
The response rate. | 24 weeks
  The response rate to treatment, defined as the percentage of patients with a decrease in HVPG of ≥10% from baseline or a decrease to below 12 mmHg after 24 weeks of treatment.
Safety assessment. | 24 weeks
  The incidence of adverse events, serious adverse events, and adverse events leading to treatment discontinuation after treatment The incidence of adverse events, serious adverse events, and adverse events leading to treatment discontinuation after treatment.

SECONDARY OUTCOMES:
Incidence of esophageal and gastric variceal bleeding during treatment. | 24 weeks
Incidence of other cirrhosis decompensation events during treatment. | 24 weeks
  other cirrhosis decompensation events: new-onset ascites/progression of ascites, spontaneous bacterial peritonitis, overt hepatic encephalopathy, acute kidney injury/hepatorenal syndrome, primary liver cancer, etc.
Degree of decrease in HVPG compared to baseline HVPG after 24 weeks of treatment. | 24 weeks
Mortality/liver transplantation rate during treatment. | 24 weeks
Overall survival time of the subjects. | 24 weeks
Degree of decrease in mean arterial pressure (MAP) compared to baseline values after treatment. | 24 weeks
Degree of decrease in heart rate compared to baseline values after treatment. | 24 weeks

OTHER OUTCOMES:
Changes in liver stiffness and spleen stiffness compared to baseline levels after 24 weeks of treatment. Changes in liver stiffness and spleen stiffness compared to baseline levels after 24 weeks of treatment. | 24 weeks
Improvement in liver function (Child-Pugh score) after 24 weeks of treatment. | 24 weeks
Improvement in liver function (MELD score) after 24 weeks of treatment. | 24 weeks
Changes in cardiac function (left ventricular ejection fraction) compared to baseline values after 24 weeks of treatment. Changes in cardiac function (left ventricular ejection fraction) compared to baseline values after 24 weeks of treatment. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Fen Xie, M.D., Principal Investigator — Shanghai Changzheng Hospital